CLINICAL TRIAL: NCT00003379
Title: A Phase I/II Study Of Whole Pelvic Radiation Therapy With Concomitant Paclitaxel and Cisplatin Chemotherapy in Patients With Cervical Carcinoma (Stages I-IV) Limited to the Pelvis
Brief Title: Radiation Therapy Plus Paclitaxel and Cisplatin in Treating Patients With Cervical Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000066374; GOG-9803
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2004-11

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; stage IB cervical cancer; stage IIB cervical cancer; stage IIA cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical small cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Paclitaxel; Brachytherapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Paclitaxel and cisplatin may increase the effectiveness of radiation therapy by making the tumor cells more sensitive to radiation. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiation therapy to the pelvis plus paclitaxel and cisplatin in treating patients who have cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of radiotherapy plus paclitaxel and cisplatin used as radiosensitization in patients with stage IB2, IIA, IIB, IIIB, or IVA invasive carcinoma of the cervix.
* Determine the maximum tolerated dose of paclitaxel when combined with cisplatin plus radiotherapy in these patients.
* Determine the effects of this regimen at the maximum tolerated dose on progression-free survival and overall survival in these patients.
* Determine the site of local or distant recurrence in these patients after treatment with this regimen.

OUTLINE: This is a dose escalation study of paclitaxel.

Patients undergo external beam radiotherapy (RT) to the pelvic region 5 days a week during weeks 1-5. Patients receive paclitaxel IV over 1 hour immediately followed by cisplatin concurrently with pelvic field radiotherapy on days 1, 8, 15, 22, 29, and 36. Patients undergo low-dose rate (LDR) OR high-dose rate (HDR) brachytherapy. For patients undergoing LDR brachytherapy, intracavitary implants are inserted 1 or 2 times within 3 weeks after completion of external beam RT. For patients undergoing HDR brachytherapy, intracavitary implants are inserted once a week for 5 weeks beginning during week 4 of external beam RT. Patients may receive a parametrial boost.

Cohorts of 3-6 patients receive escalating doses of paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued and treated at the MTD as above.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter or at time of recurrence until death.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 3-7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage IB2, IIA, IIB, IIIB, or IVA invasive carcinoma of the uterine cervix

  * Any cell type
* No metastases to para-aortic lymph nodes, scalene nodes, or to other organs outside the radiation field at time of original staging
* Study entry required within 8 weeks of diagnosis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* GOG 0-2

Life expectancy:

* More than 6 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal

Renal:

* Creatinine less than 2.0 mg/dL
* No renal abnormalities (e.g., pelvic kidney, horseshoe kidney, or renal transplantation) that would require modification of radiation fields

Other:

* Not pregnant
* No septicemia or severe infection
* No other invasive malignancy within the past 3 years except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy

Chemotherapy:

* No prior chemotherapy for this or any prior malignancy

Endocrine therapy:

* No prior endocrine therapy

Radiotherapy:

* No prior pelvic or abdominal radiotherapy for this malignancy
* No prior radiotherapy for any other prior malignancy
* No more than 1 month interval between surgery and radiotherapy

Surgery:

* See Radiotherapy

Other:

* No other prior therapy for this malignancy
* Stent or nephrostomy tube required if ureteral obstruction present

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1999-11; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan L. Walker, MD, Study Chair — Oklahoma University Cancer Institute; Michael L. Pearl, MD — Stony Brook University; Ming-teh D. Chen, MD — Women's Cancer Center - Los Gatos
Locations (31):
- United States (31):
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - Gynecologic Oncology Network, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas

REFERENCES:
- [Result] DiSilvestro PA, Walker JL, Morrison A, Rose PG, Homesley H, Warshal D; Gynecologic Oncology Group. Radiation therapy with concomitant paclitaxel and cisplatin chemotherapy in cervical carcinoma limited to the pelvis: a phase I/II study of the Gynecologic Oncology Group. Gynecol Oncol. 2006 Dec;103(3):1038-42. doi: 10.1016/j.ygyno.2006.06.017. Epub 2006 Aug 4. PMID 16889823
- [Result] Walker J, Morrison A, DiSilvestro P, et al.: GOG protocol 9803: phase I evaluation of the treatment of invasive cervical cancer confined to the pelvis with combination of radiation and weekly cisplatin and paclitaxel. [Abstract] Int J Gynecol Cancer 14 (Suppl 1): A-157, 46, 2004.